## Bringing Exposure Therapy to Real Life Context with Augmented Reality and Telepsychiatry

**Statistical Analysis Plan** 

NCT03649347

**Document Date: September 22, 2020** 

All statistical analyses will be performed in SPSS version 25 and R version 3.5.2. Data will be evaluated using standard data screening procedures. A priori power analyses were not conducted as this was a pilot study of a novel software platform; sample size was selected based on previous similar studies. Age, sex, and baseline FSQ, SPQ, and BAT will be compared between groups, in order ensure that groups do not differ at baseline. A two-way repeated measures ANOVAs will be used to measure changes in FSQ, SPQ, BAT, and CEQ over time between and within groups. The grouping variable is whether or not the individual received treatment with single-session augmented exposure. The three timepoints are baseline, one-week follow-up, and one-month follow-up. Box's M will be used to evaluate homogeneity of covariance, Levene's test will be used to evaluate homogeneity of variance, and Mauchly's Test of Sphericity will be used to evaluate sphericity. Wilk's Lambda will be the standard reported test statistic, however when any of the assumptions are violated, Pillai's Trace will be reported. For violations of sphericity, a Greenhouse-Geiser correction will be selected.